CLINICAL TRIAL: NCT05289427
Title: Triple Injection Peri-sartorius (TIPS) Block for Postoperative Analgesia After Total Knee Arthroplasty (TKA): Randomised Controlled Study
Brief Title: Triple Injection Peri-sartorius (TIPS) Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0305449
Record Dates: First submitted 2022-03-13; First posted 2022-03-21 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: Knee Disease; Nerve Pain
MeSH Terms: conditions — Neuralgia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TIPS Block (Experimental): Group TIPS; patients will receive ultrasound guided triple injection peri-sartorius block preoperatively before surgical incision
  Interventions: Procedure: ultrasound guided triple injection peri-sartorius block
- FNB (Active Comparator): Group FNB; patients will receive femoral nerve block (FNB) before surgical incision
  Interventions: Procedure: Femoral Nerve Block

INTERVENTIONS:
Procedure: ultrasound guided triple injection peri-sartorius block — Patients will receive ultrasound guided triple injection peri-sartorius block preoperatively before surgical incision
  Arms: TIPS Block
Procedure: Femoral Nerve Block — Patients will receive femoral nerve block (FNB) before surgical incision
  Arms: FNB

SUMMARY:
Comparison between the pain scores after total knee arthroplasty in patients receiving triple injection peri-sartorius (TIPS) block versus femoral nerve block (FNB)

DETAILED DESCRIPTION:
Introduction: Adequate pain control, along with quadriceps muscle preservation, has become a goal among orthopedic departments following TKA(1). The femoral nerve block (FNB) has been for many years the gold standard analgesic therapy for TKA however, it leads to quadriceps weakness(2).

Subsartorial block has been originally prescribed to block sensation in the front and the medial aspect of the knee with little quadriceps weakness (3). Local anaesthetic (LA) injected at the distal third of the adductor canal may enter into the popliteal region along with the femoral vessels to involve the popliteal plexus which supplies the posterior knee joint capsule (4). The anterior femoral cutaneous nerve (AFCN) is the overall term for the intermediate femoral cutaneous nerves (IFCNs) and the medial femoral cutaneous nerve (MFCN). The MFCN innervates the distal medial thigh as well as the anteromedial knee region. It may be anesthetized in the proximal part of the femoral triangle. The IFCN innervates the distal anterior thigh, which includes the proximal part of the surgical incision for TKA. They can be ultrasonographically identified and targeted in the subcutaneous plane on the anterior thigh where they pierce the fascia lata (FL) anterior to the sartorius muscle (SAM) before they ramify in multiple branches(5).

We hypothesize that injection of LA at the femoral triangle level above and below the sartorius muscle and at the distal end of the adductor canal may provide superior analgesia to femoral nerve block alone with little quadriceps weakness in TKA.

Aim of the study: The primary aim of this study is to compare the visual analogue scale scores during the 1st 24 postoperative hours after total knee arthroplasty in patients receiving triple injection peri-sartorius (TIPS) block versus FNB.

The secondary aims of this study are to compare the total postoperative opioid (morphine) consumption, evaluate the effect of the two techniques on the motor power of the operated limb and to detect any complications related to the block or opioids used.

Methods: After obtaining approval from Alexandria university ethics committee, this study will be carried out in El-Hadara university hospital on American Society of Anesthesiologists (ASA) physical status I-III 80 patients scheduled for unilateral TKA. A total sample size of 80 patients, 40 in each group will be sufficient to provide more than 80 % power at a two sided 0.05 significance level. The exclusion criteria will include; BMI > 35 kg/m2, pre-existing neurological deficit, any disability of the non-operated limb preventing fair mobilization, known contraindications to peripheral nerve block (coagulopathy or infection at the site of injection), or chronic opioid users/abusers.

Patients will be divided into 2 groups. Group TIPS; patients will receive ultrasound guided triple injection peri-sartorius block preoperatively before surgical incision. Group FNB; patients will receive femoral nerve block (FNB) before surgical incision.

Upon arrival to the operating room (OR), a multichannel monitor will be attached to patients, followed by the administration of 2 mg midazolam IV after securing an IV cannula. Plan of anaesthesia will be determined by the anesthesiologist in charge. After induction of general anaesthesia or administration of spinal anaesthesia, patients will be randomly divided by a closed envelope method into two groups:

Group TIPS: Patients will receive a combination of supra-sartorius plane block, femoral triangle block and distal ACB. Ten ml of 0.25 % bupivacaine will be injected. Femoral triangle block will be given just (1-2 cm) proximal to the apex of the femoral tringle which is the point at which the medial border of the sartorius muscle (STM) meets the medial border of the adductor longus muscle (ALM). Ten ml of 0.25 % bupivacaine mixed with 2 mg dexamethasone will be injected just below the STM. The needle will be withdrawn subcutaneously and another 10 ml of local anesthetic will be injected above the sartorius and below the fascia lata (5). Another 20 ml of 0.25 % bupivacaine mixed with 2 mg dexamethasone will be injected in the lower one-third of the adductor canal. At this level, femoral vessels dip into the opening of the adductor hiatus to become popliteal vessels. Sonoanatomy of this region shows the adductor magnus muscle (AMM) posteromedially, vastus medialis muscle (VMM) anterolaterally, and the STM medially.(6) Group FNB: Patients will receive single injection of 20 ml 0.25 % bupivacaine mixed with 4 mg dexamethasone about 2 cm below the inguinal ligament. LA mixture will be injected under the fascia iliaca just lateral to the femoral nerve. The femoral artery at this level will appear as a single vessel before bifurcation into profunda femoris and superficial femoral artery.

Postoperatively, multimodal analgesia regimen will be continued in the form of paracetamol 1 g /8 hours and ketorolac 30 mg /8 hours intravenously for 24 hours. Intravenous morphine at a dose of 0.05 mg/kg will be given as a rescue analgesic when the VAS ≥4. Resting and dynamic VAS assessment will be carried out every 4 hours during the 24 hour follow up period. Total postoperative morphine requirements will be measured during the postoperative follow up period.

Rehabilitation through physical therapy will be performed by patients during the 24 hour follow up period. Ambulation distances from both morning and evening sessions will be combined into a total ambulatory distance for comparative purposes. Active postoperative knee extension while patients are in seated position will be normalized into degrees of flexion (90°-0°). Physical therapy data will be obtained from physical therapy notes. Postoperative complications related to opioid usage like nausea and vomiting or related to the block like neurological symptoms or falls will be recorded. Postoperative patient satisfaction will be recorded after 24 hours.

ELIGIBILITY:
Inclusion Criteria: American Society of Anesthesiologists (ASA) physical status I-III 80 patients scheduled for unilateral total knee arthroplasty -

Exclusion Criteria:

* BMI > 35 kg/m2, Pre-existing neurological deficit, Any disability of the non-operated limb preventing fair mobilization, Known contraindications to peripheral nerve block (coagulopathy or infection at the site of injection), Chronic opioid users/abusers

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-03-07 (Actual); Study Completion 2023-03-07 (Actual)

PRIMARY OUTCOMES:
Visual Analogue scale (resting and dynamic, 11 point scale from 0 - 10 where 0 accounts for no pain and 10 accounts for worst pain) | 24 hours postoperatively
  Compare the two groups regarding the visual analogue scale scores

SECONDARY OUTCOMES:
Total postoperative morphine consumption | 24 hours postoperatively
  Compare the total postoperative opioid (morphine) consumption after total knee arthroplasty in patients receiving triple injection peri-sartorius (TIPS) block versus FNB
Operated limb motor power | 24 hours postoperatively
  Compare the two groups regarding the operated limb motor power
Complications | 24 hours
  Compare the two groups regarding complications of the two techniques and opioid related side effects

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria Faculty of Medicine, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the resultsrepoted in this article after deidentification (text, tables, figures, and appendices)
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After statistical analysis
Access Criteria: Any